CLINICAL TRIAL: NCT05167396
Title: REtinal and VIsual Cortical Response in Early PSYchosis
Acronym: REVIPSY
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Malfunctions of the Retinaute® but no adverse effects on participants. Study interrupted for BioSerenity to make technical corrections. Long immobilization of the device and conditions for reusing it not adapted to the continuation of the study.
Sponsor: Centre Psychothérapique de Nancy (Other)
Collaborators: BioSerenity (Industry); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RIPH 2021-04; n° IDRCB 2021-A01700-41 (Other: ANSM)
Record Dates: First submitted 2021-10-04; First posted 2021-12-22 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Prodromal Schizophrenia; Psychotic Episode; Prodromal Symptoms; Healthy Controls
Keywords: Electrophysiology; Vision; Retina; Visual Cortex; Early psychosis; ERG; EEG
MeSH Terms: conditions — Schizotypal Personality Disorder; Prodromal Symptoms; Psychotic Disorders

STUDY DESIGN:
Intervention Model Description: This is a cross-sectional, open, monocentric, non-randomized study applied in psychiatry and neuroscience.
  This study will include three groups of adults subject (>18 years)
  * Patients with clinical high risk of psychosis (CHRP ; n=30)
  * Patients having experienced a first psychotic episode (FEP ; n=30)
  * Healthy Controls (HC ; n=30)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Controls (HC) (Experimental): n=90
  Interventions: Device: Retinaute (BioSerenity); Device: EEG Headset 64 electrodes (BioSemi); Device: MonPackOne (Metrovision)
- Clinical High Risk of Psychosis (CHRP) (Experimental): n=30
  Interventions: Device: Retinaute (BioSerenity); Device: EEG Headset 64 electrodes (BioSemi)
- First Episode Psychosis (FEP) (Experimental): n=30
  Interventions: Device: Retinaute (BioSerenity); Device: EEG Headset 64 electrodes (BioSemi)

INTERVENTIONS:
Device: Retinaute (BioSerenity) — Wearable device in the form of a virtual reality headset for the recording of electrophysiological measurements such as electroretinogram (ERG) and electrocenphalogram (EEG), ISCEV standards
Device: EEG Headset 64 electrodes (BioSemi) — EEG headset with 64 electrodes for the recording of visual cortical electrophysiological signals
Device: MonPackOne (Metrovision) — Standard device for the recording of electroretinography (ERG) measurements, ISCEV standards
  WARNING : Device used only in 3 healthy controls to address the secondary objective
  Arms: Healthy Controls (HC)

SUMMARY:
The purpose of the REVIPSY study is to measure retinal and the visual cortical electrophysiological responses in situations at risk of psychosis in patients who have experienced a first psychotic episode. A perspective of this project will be to create new electrophysiological biomarkers predictive of the risk of conversion to psychosis

DETAILED DESCRIPTION:
The severity of psychotic disorders and their disabling potential in young patients represent a major public health problem. These populations are affected by high-level cognitive disorders associated with highly integrative functions. However, there is increasing evidence of lower-level impairments, including vision. Indeed, the literature reports electrophysiological abnormalities at the retinal level, reflected by an alteration of the signal transmission in the retinal ganglion cells (RGC), photoreceptors and bipolar cells. At the cortical level, numerous studies report electrophysiological abnormalities associated with the activity of the primary visual areas. These both electrophysiological measurements have the advantage of being objective, reliable and reproducible, thus leading to new research perspectives concerning the link between retinal and cortical measures in psychosis. These measures could also be interesting for the detection of the risk of conversion to psychosis, before it develops.

The transition to a state of psychosis is in fact marked by the appearance of symptoms, which can occur several years before the diagnosis and impact the duration of the untreated psychosis. Thus, the notion of a clinical state at high risk of psychosis (CHRP) defines a population of patients said to be at risk of psychosis. These symptoms precede the occurrence of the first psychotic episode (FEP), indicating the clear transition to psychotic illness. The questions that arise at the present time concerned the early detection and intervention of psychosis during this prodromal phase. This detection could be done via electrophysiological measures associated to the visual processing, but also via measures of neuropsychological evaluations and behavioral measures.

That is why, a study on retinal and visual cortical alterations coupled with neuropsychological assessments and behavioral measures in populations at risk of populations at risk of CHRP psychosis and in FEP would potentially reveal predictive biomarkers of the pathology. Such a project could lead to the development of retino-cortical biomarkers in mental health and will eventually lead to to create ultra-portable, reliable and routinely usable measurement devices for the early detection of psychosis in clinic.

Main objective: To measure retinal and visual cortical electrophysiological responses in clinical subjects at high risk of psychosis (CHRP) in comparison with first-episode psychotic patients (FEP) and healthy controls (CS)

Secondary objective(s) :

Compare ERG traces obtained from the "Retinaute" portable ERG device produced by the company BioSerenity with ERG traces obtained from a standard device ERG measurement device "MyPackOne" produced by the company Metrovision among healthy controls

To measure performance on neuropsychological tests in clinical subjects at high risk of psychosis (CHRP) compared to patients with a first episode of psychosis (FEP)

Measuring temporal prediction in tactile modality (unimodal) with a motor task, in clinical subjects at high risk of psychosis (CHRP) in comparison with first-episode patients (FEP) and healthy controls (CS)

Measuring temporal prediction in visual and tactile (multimodal) modalities/Measuring temporal prediction in visual modality (unimodal) with a classical perceptual task in clinical subjects at high risk of psychosis (CHRP) in comparison with patients with a first psychotic episode with a first episode of psychosis (FEP) and healthy controls (CS)

To compare the sensitivity of behavioural and EEG measures to the prediction of tactile vs. visual stimuli, and multimodal vs. unimodal

ELIGIBILITY:
1. Inclusion Criteria:

   1. All groups

      Age and gender matching

      Age between 18 and 40

      Enrolled in a social security plan

      Normal or corrected-to-normal visual acuity verified by Monoyer test

      In women of childbearing age: negative urine pregnancy test at the inclusion visit

      Person who has received and understood prior information about the study

      Person who has given free and informed written consent prior to any participation in the study
   2. Healthy control group (HC; n=30)

      Met "all groups" criteria

      No current disorders as assessed by the MINI global assessment

      No lifetime (hypo)manic episodes or psychotic disorders and current

      No current or past disorders by CAARMS assessment

      No current disorders according to ICD-10 criteria

      No positive family history (parents/first degree) for affective affective, non-affective psychoses or major affective disorders

      No regular use (more than 3 psychotropic medications: benzodiazepines, hypnotics,antidepressants, antipsychotics or mood regulators or psychostimulants) during the past last 12 months
   3. High clinical risk group for psychosis (CHRP; n=30)

      Met "all groups" criteria, Assessment at CAARMS:
      * Attenuated positive symptoms (APS)
      * OR Brief Intermittent Psychotic Symptoms (BIPS)
      * OR Attenuated psychosis of sub-laminar frequency
      * OR sub-laminar attenuated psychosis

      Antipsychotic treatment with a cumulative dose of equivalent chlorpromazine <2500mg lifetime (1)
   4. First Episode Psychosis (FEP; n=30)

   All-group criteria met CAARMS assessment: Psychosis/antipsychotic treatment threshold treatment threshold achieved at CAARMS

   Antipsychotic treatment with a cumulative dose of equivalent chlorpromazine <2500mg lifetime (1)
2. Exclusion Criteria (all groups):

Impairment of the subject that makes it difficult or impossible to participate in the or comprehension of the information provided to him/her

Dyslexia

Substance use disorder according to CIM-10

Neurological history including progressive neurological pathology

Progressive retinal disease

Chronic glaucoma

Ophthalmologic pathology affecting visual acuity

Current ocular infection

Major under guardianship, curatorship or safeguard of justice

Pregnant or breastfeeding women

Persons in a life-threatening emergency situation

Result of the preliminary medical examination incompatible with the research

Patient presenting a suicidal risk.

Criteria incompatible with the use of the Retinaute:

* Allergy to silver
* Known or suspected allergy to any of the following components:

polyamide, polyester, elastane, latex, rubber, silicone, or any synthetic material as well as to cotton in case the device is used without the device is used without a protective head covering

* Sensory disorders making the patient insensitive to pain on the skin.
* Behavioral problems making the patient extremely agitation or aggression.
* Mental disorders incompatible with the use of the device.
* Seizure disorder.
* Open wound in an area covered or wrapped by the device.
* User at high risk of contagion.
* Wearing an implantable medical device (e.g. pacemaker)
* Pregnant women, women in labor or nursing mothers.
* Allergy or skin sensitivity to one of the components of the cream Elefix or equivalent on the market: coconut oil, egg oil, propylene glycol egg oil, propylene glycol, glycerin, lanolin...
* Allergy or skin sensitivity to one of the components of the cream NuPrep or market equivalent

Participation in another interventional study (exclusion period included)

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-01-26 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
N95 wave | Day1
  Amplitude
a wave | Day1
  Amplitude
b wave | Day1
  Amplitude
P100 wave | Day1
  Amplitude

SECONDARY OUTCOMES:
Visual Object and Space Perception (VOSP) | Day1
  Score
Verbal Fluency | Day1
  Score
Working Memory | Day1
  Score
Betarythm (EEG oscillatory responses) | Day1
  Amplitude
Contingent Negative Variation (CNV) | Day1
  Amplitude reaction time between a warning and a go signal as measured by electroencephalography (EEG)
CPT-AX (Continuous Performance Task version AX) | Day1
  Score
fNART (French adaptation of National Adult Reading Test) | Day1
  Score
TAP (Test of Attentional Performance) | Day1
  Score

CONTACTS AND LOCATIONS:
Overall Officials: Vincent LAPRÉVOTE, Pr. MD PhD, Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Centre Psychothérapeutique de Nancy, Laxou, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laprevote V, Heitz U, Di Patrizio P, Studerus E, Ligier F, Schwitzer T, Schwan R, Riecher-Rossler A. [Why and how to treat psychosis earlier?]. Presse Med. 2016 Nov;45(11):992-1000. doi: 10.1016/j.lpm.2016.07.011. Epub 2016 Aug 21. French. PMID 27554461
- [Background] Demmin DL, Davis Q, Roche M, Silverstein SM. Electroretinographic anomalies in schizophrenia. J Abnorm Psychol. 2018 May;127(4):417-428. doi: 10.1037/abn0000347. PMID 29745706
- [Background] Moghimi P, Torres Jimenez N, McLoon LK, Netoff TI, Lee MS, MacDonald A 3rd, Miller RF. Electoretinographic evidence of retinal ganglion cell-dependent function in schizophrenia. Schizophr Res. 2020 May;219:34-46. doi: 10.1016/j.schres.2019.09.005. Epub 2019 Oct 12. PMID 31615740
- [Background] Tan A, Schwitzer T, Conart JB, Angioi-Duprez K. [Retinal investigations in patients with major depressive disorder, bipolar disorder or schizophrenia: A review of the literature]. J Fr Ophtalmol. 2020 Sep;43(7):586-597. doi: 10.1016/j.jfo.2019.10.029. Epub 2020 Jul 4. French. PMID 32631695
- [Background] Butler PD, Martinez A, Foxe JJ, Kim D, Zemon V, Silipo G, Mahoney J, Shpaner M, Jalbrzikowski M, Javitt DC. Subcortical visual dysfunction in schizophrenia drives secondary cortical impairments. Brain. 2007 Feb;130(Pt 2):417-30. doi: 10.1093/brain/awl233. Epub 2006 Sep 19. PMID 16984902
- [Background] Knebel JF, Javitt DC, Murray MM. Impaired early visual response modulations to spatial information in chronic schizophrenia. Psychiatry Res. 2011 Sep 30;193(3):168-76. doi: 10.1016/j.pscychresns.2011.02.006. Epub 2011 Jul 20. PMID 21764264
- [Background] Kim DW, Shim M, Song MJ, Im CH, Lee SH. Early visual processing deficits in patients with schizophrenia during spatial frequency-dependent facial affect processing. Schizophr Res. 2015 Feb;161(2-3):314-21. doi: 10.1016/j.schres.2014.12.020. Epub 2014 Dec 29. PMID 25553978